CLINICAL TRIAL: NCT04720729
Title: Chemotherapy Monitoring by Circulating Tumor DNA (ctDNA) in HER2 (Human Epidermal Growth Factor Receptor-2)- Metastatic Breast Cancer (MONDRIAN): a Phase 2 Study
Brief Title: Chemotherapy Monitoring by ctDNA in HER2- Metastatic Breast Cancer
Acronym: MONDRIAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2020-10
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: HER2-negative Metastatic Breast Cancer

STUDY DESIGN:
Intervention Model Description: Single arm phase 2 study, Chemotherapy monitoring based on ctDNA early changes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients with HER2-negative metastatic breast cancer, starting a second line of chemotherapy
  Interventions: Biological: Chemotherapy monitoring by circulating tumor DNA analysis

INTERVENTIONS:
Biological: Chemotherapy monitoring by circulating tumor DNA analysis — During the screening step (2nd chemotherapy line, cycle 1) : at each time point (L2C1D1 & L2C1D15), 30 ml of blood will be drawn on special tubes with conservative suited for ctDNA analyses (e.g. STRECK® tubes).Then cell-free circulating DNA (cfcDNA) will be extracted from plasma following the manufacturer recommendations. cfcDNA will be quantified, and minimum 500-1000 copies will be analyzed by droplet digital PCR (ddPCR). Analyses will define if ctDNA could be detected during L2.
  For the interventional step, from L3 (3rd chemotherapy line) : 20 ml of blood will be drawn at L3C1D1 and L3C1D15. If ctDNA at D15 shows a major drop (> 40%) from D1, treatment will be continued. If ctDNA at D15 shows no major drop from D1, chemotherapy will be changed.

SUMMARY:
This is a one-arm, single site, open-label phase II study. Patients will be enrolled in the screening step at the start of the second line of chemotherapy, and will undergo blood draws for ctDNA detection. Patients for whom ctDNA was successfully detected and found informative by the study executive board could then be included in the interventional step when starting a new line of therapy.

ctDNA will be quantified using the customized test, at baseline and day 15 (+/- 3 working day) of cycle #1, and results will be made available before the cycle 2 Day 1, together with a treatment management recommendation by the Study Executive Board (continuation or discontinuation of the corresponding chemotherapy)

DETAILED DESCRIPTION:
Patients will be enrolled in the screening step at the start of the second line of chemotherapy, and will undergo blood draws for ctDNA detection:

That second line of treatment will be managed by clinical and radiological evaluations (RECIST); ctDNA will not be released to clinician and patient in real time.

While the included patient is being treated by second line therapy, a customized ctDNA detection based on tumor mutations (droplet-digital PCR) will be developed. Once set up, the two blood above-mentioned samples will be subjected to ctDNA detection. The SEB will then retrospectively assess whether ctDNA levels changes during the second line of treatment were indicative of the efficacy of the second line therapy. Patients for whom ctDNA was successfully detected and found informative by the SEB (Steering Executive Board) could then be included in the interventional step when starting a new line of therapy.

The third blood draw for ctDNA detection will be used to compare results to the tumor evaluation performed by imaging.

In the interventional step, ctDNA analyses and interpretation will be performed in real time; results made available before the cycle 2. Quantitative results will be interpreted by the laboratory committee, with two possible recommendations:

* ctDNA changes at day 15 display a major drop (Mutant Allelic Frequency (MAF) or copies/ml) reduced by 40% or more compared to baseline: continuing the same chemotherapy will be recommended;
* ctDNA changes at day 15 display no major drop (MAF or copies/ml) either increased, stable or reduced by less than 40% compared to baseline: changing chemotherapy will be recommended; In light of ctDNA levels changes observed during the second line for each included patient, the above-mentioned thresholds might be modified, on a case-by-case basis, by the SEB (to keep into account individual characteristics).

The test will be repeated for any new line of therapy that may be initiated during the first 6 months following the accrual of each patient in the interventional step. If this strategy is considered efficient (on an individual basis), further ctDNA tests will be made available on request for the next six months. Consequently, the patients who will change chemotherapy line after the recommendation following result from C1D15 ctDNA results will have a new ctDNA test at C1D1 and C1D15 of the new chemotherapy line.

ELIGIBILITY:
Inclusion criteria :

* Written informed consent
* Woman ≥ 18 years old
* Performance status 0-2
* Advanced HER2-negative metastatic breast cancer on the last tumor tissue assessed (ASCO-CAP (College of American Pathologists) guidelines)
* Eligible to a second line of chemotherapy for MBC (Metastatic Breast Cancer)
* Evaluable disease (per RECIST v1.1)
* Organ functions compatible with the use of chemotherapies (as decided by the investigator)
* No isolated CNS progression or leptomeningeal carcinomatosis
* No concurrent stage IV malignancy
* No concurrent severe and/or uncontrolled medical or psychological condition that would contraindicate participation in this study

Additional criteria for the screening step :

Presence of a known somatic mutation deemed trackable in circulating cell-free DNA. If the tumoral genetic landscape is unknown at inclusion, its characterization should be requested (or ongoing) at inclusion

Additional criteria for the interventional step :

* Satisfactory ctDNA detection and changes during the 2nd line, as determined by the Study Executive Board (SEB)
* Patient eligible to a third line of chemotherapy

Exclusion criteria :

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer,
Enrollment: 160 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
L3C1 : ctDNA quantification | At the Day 1 of Cycle 1 (each cycle is 21 days)
  ctDNA quantification (Mutant Allelic Frequency (MAF) %) during 3rd chemotherapy Line, 1st cycle (L3C1)
L3C1 : ctDNA quantification | At the Day 15 of Cycle 1 (each cycle is 21 days)
  ctDNA quantification (Mutant Allelic Frequency (MAF) %) during 3rd chemotherapy Line, 1st cycle (L3C1)
L3C1 : chemotherapy efficacy | ctDNA difference between Day 15 and Day 1
  ctDNA change : if major drop from D1 to D15 (MAF>40%), no change on treatment. If no major drop from D1 to D15, change of chemotherapy
LxC1 : ctDNA quantification | At the Day 1 of the Cycle 1 (each cycle is 21 days)
  ctDNA quantification (MAF %) during 4th chemotherapy line and following : Line x, 1st cycle (LxC1)
LxC1 : ctDNA quantification | At the Day 15 of the Cycle 1 (each cycle is 21 days)
  ctDNA quantification (MAF %) during 4th chemotherapy line and following : Line x, 1st cycle (LxC1)
LxC1 : chemotherapy efficacy | ctDNA difference between Day 15 and Day 1
  ctDNA change : if major drop from D1 to D15 (MAF>40%), no change on treatment recommanded If no major drop from D1 to D15, change of chemotherapy recommanded
Progression Free Survival (PFS) | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed every 8-weeks up to 18 months
  Tumor assessment (MRI and/or CT) by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, PR, Study Director — INSTITUT CURIE - Medical Oncology; Steven LE GOUILL, PR, MD, Study Chair — INSTITUT CURIE - Hospital
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No